CLINICAL TRIAL: NCT03541174
Title: Multi-center, Blinded, Randomized, Parallel-group, Phase 3 Study With Aprocitentan in Subjects With Resistant Hypertension (RHT)
Brief Title: A Research Study to Show the Effect of Aprocitentan in the Treatment of Difficult to Control (Resistant) High Blood Pressure (Hypertension) and Find Out More About Its Safety
Acronym: PRECISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-080A301; 2017-004393-33 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Resistant Hypertension
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Intervention Model Description: Study with multiple periods and parts.
  Once eligibility is confirmed during screening and the run-in period, the individuals entered the randomized treatment period consisting of 3 parts: Part 1: double-blind (DB), randomized to aprocitentan 12.5 mg, aprocitentan 25 mg or placebo; Part 2 single-blind (SB) aprocitentan 25 mg; Part 3: double-blind withdrawal (DB-WD) re-randomized to aprocitentan 25 mg or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Aprocitentan 25 mg in Part 1 (double-blind) (Experimental): Participants will receive aprocitentan 25 mg, orally, once daily in the morning for 4 weeks.
  Interventions: Drug: Aprocitentan 25 mg
- Aprocitentan 12.5 mg in Part 1 (double-blind) (Experimental): Participants will receive aprocitentan 12.5 mg, orally, once daily in the morning for 4 weeks.
  Interventions: Drug: Aprocitentan 12.5 mg
- Placebo in Part 1 (double-blind) (Placebo Comparator): Participants will receive placebo (matching aprocitentan), orally, once daily in the morning for 4 weeks.
  Interventions: Drug: Placebo
- Aprocitentan 25 mg in Part 2 (single-blind, single arm) (Experimental): After 4-weeks in the double-blind randomized part (Part 1), participants will received 25 mg aprocitentan, orally, once daily in the morning for 32 weeks.
  Interventions: Drug: Aprocitentan 25 mg
- Aprocitentan 25 mg in Part 3 (double-blind withdrawal) (Experimental): After 32-weeks in the single-blind, single-arm part (Part 2), participants will be re-randomized and receive aprocitentan 25 mg, orally, once daily in the morning for 12 weeks.
  Interventions: Drug: Aprocitentan 25 mg
- Placebo in Part 3 (double-blind withdrawal) (Placebo Comparator): After 32-weeks in the single-blind, single-arm part (Part 2), participants will be re-randomized and receive placebo (matching aprocitentan), orally, once daily in the morning for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprocitentan 12.5 mg — Tablet, oral use
  Other Names: ACT-132577
  Arms: Aprocitentan 12.5 mg in Part 1 (double-blind)
Drug: Aprocitentan 25 mg — Tablet, oral use
  Other Names: ACT-132577
  Arms: Aprocitentan 25 mg in Part 1 (double-blind); Aprocitentan 25 mg in Part 2 (single-blind, single arm); Aprocitentan 25 mg in Part 3 (double-blind withdrawal)
Drug: Placebo — Matching placebo tablet
  Arms: Placebo in Part 1 (double-blind); Placebo in Part 3 (double-blind withdrawal)

SUMMARY:
The goal of this clinical trial is to show the blood pressure lowering effect of aprocitentan, a new drug, when added to other anti-hypertensive drugs of patients with difficult to control (resistant) high blood pressure (hypertension), and to show that blood pressure reduction is kept for long period of time.

DETAILED DESCRIPTION:
Participation in the study will be up to 68 weeks.

The study has 4 periods:

1. Screening period
2. Placebo run-in period
3. Randomized treatment period
4. Safety follow-up period

The screening period lasts between 4 and 12 weeks. It starts at the screening visit with the signing of the informed consent form (ICF) and ends the day before the participant enters the run-in period.

At least 4 weeks before the start of the run-in period, the background antihypertensive medication (except beta-blockers) of participants with a diagnosis of true resistant hypertension and having a mean trough sitting systolic blood pressure of equal to or greater than 140 mmHg measured by automated AOBPM will be standardized by switching to a fixed combination of a calcium channel blocker (amlodipine), an angiotensin receptor blocker (valsartan) and a diuretic (hydrochlorothiazide).

In case a beta-blocker is used as one of the background antihypertensive medications or for any other indication, this can be kept, with the provision that it has been initiated and the dose kept stable for at least 4 weeks prior to the screening visit and the dose kept stable until the end-of-treatment.

Following the screening period this study has a run-in period of 4 weeks. During this period, placebo will be administered in order to exclude potential placebo responders.

Following the run-in period eligible participants will enter the randomized treatment period. This period lasts for 48 weeks. It starts at randomization (i.e., Day 1 of the double-blind part) and ends at the end-of-treatment visit (i.e., at the end of the double-blind withdrawal part).

The randomized treatment period consists of 3 parts: Part 1 is double-blind, randomized, parallel-group and placebo-controlled and lasts 4 weeks. Part 2 is single-blind and single-arm and lasts for 32 weeks. Part 3 is a double-blind withdrawal, randomized, parallel-group and placebo-controlled and lasts for 12 weeks.

End-of treatment is at Week 48 (i.e., end of the double-blind withdrawal part). The safety follow-up starts on the day after the last dose of study treatment and ends 30 to 33 days after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

Screening period:

* Signed and dated informed consent form (ICF) prior to any study-mandated procedure;
* Male and female participants; 18 years (or year of country specific majority) or older;
* Historical documentation in the participant's medical records on uncontrolled blood pressure despite at least 3 background antihypertensive medications within 1 year before screening visit;
* Treated with at least 3 antihypertensive therapies of different pharmacological classes for at least 4 weeks before the screening visit (Visit 1);
* Mean Sitting Systolic Blood Pressure (SiSBP) greater or equal to 140 mmHg measured by Automated Office Blood Pressure Measurement (AOBPM);
* Women of childbearing potential are eligible only if the following applies:

  * Negative pregnancy test at screening and at baseline (i.e., before randomization);
  * Agreement to undertake pregnancy tests during the study and up to 30 days after randomized study treatment discontinuation;
  * Agreement to use methods of birth control from Screening up to at least 30 days after randomized study treatment discontinuation.

Run-in period (RI):

* Switched to the standardized background antihypertensive therapy at least 4 weeks before the first RI visit;
* Mean trough SiSBP greater than or equal to140 mmHg as measured by AOBPM.

Randomization period:

* Stable dose of the standardized background antihypertensive therapy for at least 1 week before the end of the RI period;
* Mean trough SiSBP greater than or equal to 140 mmHg measured by AOBPM.

Exclusion Criteria:

* Apparent/pseudo Resistant Hypertension (RHT) due to white coat effect, medical inertia, poor therapeutic adherence, or secondary causes of hypertension (except sleep apnea);
* Confirmed severe hypertension (grade 3) defined as SiSBP greater than or equal to 180 mmHg and/or Sitting Diastolic Blood Pressure (SiDBP) greater than or equal to 110 mmHg as measured by AOBPM at two different timepoints;
* Pregnant or lactating participants;
* Clinically significant unstable cardiac disease at screening or in the past in the opinion of the investigator (exclusion of participants with significant or potential unstable cardiac disease);
* Severe renal insufficiency;
* Any known factor, disease or clinically relevant medical or surgical conditions that, in the opinion of the investigator, might put the participant at risk, interfere with treatment compliance, study conduct or interpretation of the results.
* Treatment with any medication which may affect blood pressure (BP) and/or treatment with high dose of loop diuretics (i.e., furosemide greater than 80 mg/day, or equivalent dosage of other loop diuretics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (159):
- United States (41):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Chrishard Medical Group, Inglewood, California
  - Clinical Trials Research, Lincoln, California
  - Academic Medical Research Institute Inc, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - California Kidney Specialists, San Dimas, California
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Century Clinical Research, Inc, Daytona Beach, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Canvas Clinical Research, LLC, Lake Worth, Florida
  - East Coast Institute for Research, Saint Augustine, Florida
  - Premier Medical Associates, The Villages, Florida
  - SIU School of Medicine Center for Clinical Research, Springfield, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana, L.L.C., Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Grace Research, LLC, Bossier City, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Hypertension and Nephrology Association PA, Eatontown, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Scott Research Inc, Laurelton, New York
  - Great Lakes Medical Research LLC, Westfield, New York
  - Metrolina Internal Medicine/Internal Medicine Research, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - University Hospitals Cleveland Medical Center - Neurological Institute, Cleveland, Ohio
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - TLM Medical Services LLC, Columbia, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - LifeDOC Research PLLC, Memphis, Tennessee
  - Amarillo Heart Clinical Research Institute, Inc., Amarillo, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Mercury Clinical Research, Webster, Texas
  - St. George Kidney Care LLC dba Southern Utah Kidney and Hypertension Center, St. George, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Milwaukee Nephrologists, SC, Wauwatosa, Wisconsin
- Australia (6):
  - Renal Research, Gosford, New South Wales
  - Westmead Hospital Department of Renal Medicine, Sydney, New South Wales
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - Hypertension & Kidney Disease / Huma Neurotransmitter Laboratory, Melbourne, Victoria
  - Curtin University, Faculty of Health Sciences, School of Public Health, Bentley, Western Australia
  - Royal Perth Hospital Unit - The University of Western Australia, Perth, Western Australia
- Belgium (4):
  - Hospital Erasme - Cardiology department, Brussels
  - Clinique Universitaires de Saint Luc, Departement cardio-vasculaires intensives, Brussels
  - Universitair Ziekenhuis Gent Cardiologie, Ghent
  - Centre Hospitalier Universitaire du Sart-Tilman, Liège
- Canada (5):
  - Manna Research Inc (North Burlington), Hamilton, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Stephen S. Chow Medicine Professional Corporation, Toronto, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
- China (7):
  - The First Affiliated Hospital of Baotou Medical College of Inner Mongolia, Baotou
  - The Third Xiangya Hospital of Central South University, Changsha
  - Guangdong General Hospital, Guangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - Hainan NO.3 Provincial people's Hospital, Sanya
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- Czechia (5):
  - FN U Sv.Anny Brno, kardiologická klinika, Brno
  - Všeobecní fakultní nemocnice Praha, Prague
  - Thomayerova nemocnice, Prague
  - Interni oddeleni, Nefrologie, Prague
  - Kardio Václavík s.r.o, Přerov
- Finland (3):
  - University of Oulu, Medical Research Center, Oulu
  - TAYS RDI center (Tampere University Hospital,Specialist Internal Medicine, Rare Diseases), Tampere
  - Turku University Central Hospital - Turun yliopistollinen keskussairaala Sisätautien klinikka, Turku
- France (4):
  - CHU Grenoble - Alpes, Grenoble
  - Hôpital de la Croix-Rousse - Rhône, Lyon
  - Hôpital Européen Georges Pompidou- Centre d' Investigation Clinique, Paris
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon
- Germany (6):
  - Jewish Hospital Berlin, Berlin
  - Universitätsklinikum Düsseldorf Klinik für Nephrologie, Düsseldorf
  - Universitätsklinikum Erlangen Klinische Forschungsstation (CRC), Erlangen
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Herzzentrum Leipzig Universitätsklinik für Kardiologie, Leipzig
  - Universitätsklinikum Nürnberg Süd, Nuremberg
- Greece (4):
  - General Hospital of Athens, Ippokrateio, Athens
  - General Hospital of Athens Georgios Gennimatas, Athens
  - Asklepeion General Hospital, Athens
  - General Hospital Konstantopouleio-Patision, Nea Ionia
- Hungary (4):
  - DRC Gyógyszervizsgáló Központ Kft., Balatonfüred
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Debreceni Egyetem - Klinikai Központ, Debrecen
  - Markusovszky Egyetemi Oktatókórház, Szombathely
- Israel (5):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Cardiovascular Institute, Ashkelon
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - University Brescia Department Clinical and Experimental Science, Brescia
  - Ospedale San Gerardo, Clinica Medica, Monza
  - Azienda Ospedaliero Universitaria Pisana - Department Clinical and Experimental Medicine, Pisa
  - Azienda Ospedaliera S. Andrea di Roma - Division of Cardiology and of Cardiothoracic and Vascular Science Department -, Roma
  - SCU Medicina Interna e Centro Ipertensione arteriosa. Dipartimento di Scienze Mediche Università di Torino, Aou Citta' Salute E Scienza Torino, Torino
- Lithuania (2):
  - JSC "InMedica", Kaunas
  - Clinic of Cardiology and Rehabilitation, Klaipėda
- Netherlands (4):
  - Academic Medical Center Amsterdam, Amsterdam
  - Zuyderland Medical Center, Geleen
  - Maastricht University Medical Center, Dept. of Medicine, Maastricht
  - Radboud University Medical Center, Nijmegen
- Poland (15):
  - Uniwersyteckie Centrum Kliniczne Centrum Kardiologii, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mielęckiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Diamond Clinic, Krakow
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - KO-MED. CentraKliniczne Sp. Z o.o. Ośrodek Badań Klinicznych w Lublinie II, Lublin
  - ETG Lublin, Lublin
  - Etyka Ośrodek Badań Klinicznych, Olsztyn
  - KO-MED. Centra Kliniczne Sp. Z o.o. Ośrodek Badań Klinicznych w Puławach, Puławy
  - ETG Skierniewice, Skierniewice
  - Medycyna Kliniczna, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
  - ETG Warszawa, Warsaw
  - Klinika Wad Wrodzonych Serca Instytut Kardiologii im. Kardynala Wyszynskiego, Warsaw
  - Samodzielny Publiczny Szpital Wojewódzki im. Papieża Jana Pawła II w Zamościu, Zamość
  - ETG Zgierz, Zgierz
- Russia (15):
  - State Budgetary Healthcare Institution of Arkhangelsk Region "First City Clinical Hospital n.a. E.E. Volosevich", Arkhangelsk
  - Federal State Autonomous Institution of Higher Education "Kazan (Volga Region) Federal University", Kazan'
  - Federal State Budget Scientific Institution "Scientific Research Institute for Complex Issues of Cardiovascular Diseases", Kemerovo
  - Scientific Research Institute - Regional Clinical Hospital №1, Krasnodar
  - National Medical Research Center for Preventive Medicine, Moscow
  - State budget healthcare institution of Novosibirsk region "City clinical hospital #34", Novosibirsk
  - Federal State Budget Scientific Institution "Federal Research Center Institute of Cytology and Genetics of Siberian Department of Russian Academy of Sciences", Novosibirsk
  - Federal State Military Educational Institution of Higher Professional Education, Military Medical Academy named for S. M. Kirov of the Ministry of Defense of the Russian Federation, Saint Petersburg
  - Federal State Budget Institution "National Medical Research Center n.a. V.A. Almazov" of the Ministry of healthcare of the Russian Federation, Saint Petersburg
  - Federal State Budget Institution National Medical Research Center n.a. V.A. Almazov of the Ministry of Healthcare of the Russia, Saint Petersburg
  - State Healthcare Institution "Regional Clinical Cardiology Dispensary", Saratov
  - Federal State Budget Educational Institution of Higher Education "Saratov State Medical University n.a. V.I. Razumovskiy" of the Ministry of Healthcare of the Russian Federation, Saratov
  - State Budgetary Educational Institution of Higher Professional Education Smolensk State Medical Academy, Smolensk
  - Federal State Budget Scientific Institution "Tomsk National Research Medical Center of the Russian Academy of Sciences", Tomsk
  - Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen
- Spain (10):
  - Hospital del Mar, Barcelona
  - Fundació Puigvert, Barcelona
  - Hospital Vall d'Hebron de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Virgen de las Nieves - Internal Medicine Department, Granada
  - Hospital Clinico San Carlos - Istituto de Investigacion Sanitaria San Carlos (IdISSC), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Rocio Departamento de Medicina Interna, Seville
  - Hospital Clínic Universitari de València, Valencia
  - Hypertension Clinic, Internal Medicine, Hospital Clinico, University of Valencia, Valencia, Valencia
- Ukraine (11):
  - State Institution "L.T. Malaya Therapy National Institute of the NAMS of Ukraine", Kharkiv
  - Municipal non-profit enterprise "Clinical Hospital # 8"of Kharkiv City Council, Kharkiv
  - Kyiv City Clinical Hospital # 1, Kyiv
  - Kyiv Municipal Clinical Emergency Hospital, Kyiv
  - State Institution "National Scientific Center "M.D. Strazhesko Institute of Cardiology" of the National Academy of Medical Sciences of Ukraine", Kyiv
  - State Institution "D.F. Chebotarev Institute of Gerontology, National Academy of Medical Science of Ukraine", Kyiv
  - State Institution "Institute of Gerontology named after D.F. Chebotarev of National Academy of Medical Sciences of Ukraine", Kyiv
  - Volyn Regional Center for Cardiovascular Pathology, Rehabilitation Department, Lutsk
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Communal Non-profit Enterprise "Vinnytsya regional Clinical Hospital named after. N.I. Pirogov Vinnytsia Regional Council"/ National Pirogov Memorial Medical University, Vinnytsya, Vinnytsia
  - O.F. Herbachevsky Zhytomyr Regional Clinical Hospital, Cardiology department, Zhytomyr
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Clinical Pharmacology Unit, Aberdeen
  - Clinical Research Centre The University of Edinburgh Centre for Cardiovascular Science, Edinburgh
  - Queen Mary University of London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daskalopoulou SS, Khan NA, Quinn RR, Ruzicka M, McKay DW, Hackam DG, Rabkin SW, Rabi DM, Gilbert RE, Padwal RS, Dawes M, Touyz RM, Campbell TS, Cloutier L, Grover S, Honos G, Herman RJ, Schiffrin EL, Bolli P, Wilson T, Feldman RD, Lindsay MP, Hemmelgarn BR, Hill MD, Gelfer M, Burns KD, Vallee M, Prasad GV, Lebel M, McLean D, Arnold JM, Moe GW, Howlett JG, Boulanger JM, Larochelle P, Leiter LA, Jones C, Ogilvie RI, Woo V, Kaczorowski J, Trudeau L, Bacon SL, Petrella RJ, Milot A, Stone JA, Drouin D, Lamarre-Cliche M, Godwin M, Tremblay G, Hamet P, Fodor G, Carruthers SG, Pylypchuk G, Burgess E, Lewanczuk R, Dresser GK, Penner B, Hegele RA, McFarlane PA, Sharma M, Campbell NR, Reid D, Poirier L, Tobe SW; Canadian Hypertension Education Program. The 2012 Canadian hypertension education program recommendations for the management of hypertension: blood pressure measurement, diagnosis, assessment of risk, and therapy. Can J Cardiol. 2012 May;28(3):270-87. doi: 10.1016/j.cjca.2012.02.018. PMID 22595447
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Result] Danaietash P, Verweij P, Wang JG, Dresser G, Kantola I, Lawrence MK, Narkiewicz K, Schlaich M, Bellet M; PRECISION investigators. Identifying and treating resistant hypertension in PRECISION: A randomized long-term clinical trial with aprocitentan. J Clin Hypertens (Greenwich). 2022 Jul;24(7):804-813. doi: 10.1111/jch.14517. Epub 2022 Jun 9. PMID 35686330
- [Derived] Rossignol P, Clozel M, Dreier RF, Flack JM, Flamion B, Mann J, Narkiewicz K, Sassi-Sayadi M, Wang JG, Weber MA, Schlaich MP. Aprocitentan in Patients With Chronic Kidney Disease and Resistant Hypertension. Hypertension. 2026 Feb;83(2):e25563. doi: 10.1161/HYPERTENSIONAHA.125.25563. Epub 2025 Dec 9. PMID 41363010
- [Derived] Flack JM, Schlaich MP, Weber MA, Sassi-Sayadi M, Narkiewicz K, Clozel M, Dreier RF, Andrawis NS, Danaietash P, Gabra N, Scott D, Wang JG, Ferdinand KC. Aprocitentan for Blood Pressure Reduction in Black Patients. Hypertension. 2025 Apr;82(4):601-610. doi: 10.1161/HYPERTENSIONAHA.124.24142. Epub 2025 Jan 22. PMID 39840441
- [Derived] Xu J, Jiang X, Xu S. Aprocitentan, a dual endothelin-1 (ET-1) antagonist for treating resistant hypertension: Mechanism of action and therapeutic potential. Drug Discov Today. 2023 Nov;28(11):103788. doi: 10.1016/j.drudis.2023.103788. Epub 2023 Sep 22. PMID 37742911
- [Derived] Schlaich MP, Bellet M, Weber MA, Danaietash P, Bakris GL, Flack JM, Dreier RF, Sassi-Sayadi M, Haskell LP, Narkiewicz K, Wang JG; PRECISION investigators. Dual endothelin antagonist aprocitentan for resistant hypertension (PRECISION): a multicentre, blinded, randomised, parallel-group, phase 3 trial. Lancet. 2022 Dec 3;400(10367):1927-1937. doi: 10.1016/S0140-6736(22)02034-7. Epub 2022 Nov 7. PMID 36356632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was done from 18 June 2018 to 25 April 2022.
Pre-assignment Details: 730 participants are considered to be enrolled in the study and were randomized to study treatment.
Groups:
- Aprocitentan 12.5 mg in Part 1 (Double-blind): Participants were randomized and received aprocitentan 12.5 mg, orally, once daily in the morning for 4 weeks.
- Aprocitentan 25 mg in Part 1 (Double-blind): Participants were randomized and received aprocitentan 25 mg, orally, once daily in the morning for 4 weeks.
- Placebo in Part 1 (Double-blind): Participants were randomized and received placebo (matching aprocitentan), orally, once daily in the morning for 4 weeks.
- Aprocitentan 25 mg in Part 2 (Single-blind): Participants that completed the double-blind part received aprocitentan 25 mg, orally, once daily in the morning for 32 weeks.
- Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal): After the 32-week single-blind, single-arm aprocitentan 25 mg (Part 2), participants were re-randomized and received aprocitentan 25 mg, orally, once daily in the morning for 12 weeks.
- Placebo in Part 3 (Double-blind Withdrawal): After the 32-week single-blind, single-arm aprocitentan 25 mg (Part 2), participants were re-randomized and received placebo (matching aprocitentan), orally, once daily in the morning for 12 weeks.
Period: Part 1 Double-Blind
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 2 (Single-blind) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Started | 243 | 243 | 244 | 0 | 0 | 0
Safety Set (Two participants randomized to placebo received at least one dose of aprocitentan 25 mg during double-blind part 1.) | 243 | 245 | 242 | 0 | 0 | 0
Completed | 232 | 234 | 238 | 0 | 0 | 0
Not Completed | 11 | 9 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 5 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Other reasons | 3 | 2 | 3 | 0 | 0 | 0
Period: Part 2 Single-Blind
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 2 (Single-blind) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Started | 0 (The 232 participants that completed 12.5 mg aprocitentan study treatment in part 1 entered the single-blind 25 mg aprocitentan arm in part 2.) | 0 (The 236 participants that completed 25 mg aprocitentan study treatment in part 1 entered the single-blind 25 mg aprocitentan arm in part 2.) | 0 (The 236 participants that completed placebo study treatment in part 1 entered the single-blind 25 mg aprocitentan arm in part 2.) | 704 (Total number of participants that completed the double-blind part 1 who entered the single-blind, single-arm part 2.) | 0 | 0
Completed | 0 | 0 | 0 | 613 | 0 | 0
Not Completed | 0 | 0 | 0 | 91 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 25 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 19 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 8 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 32 | 0 | 0
Period: Part 3 Double-Blind Withdrawal
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 2 (Single-blind) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Started | 0 | 0 | 0 | 0 | 307 | 307
Safety Set (613 participants started study treatment in Part 3. Four participants re-randomised to placebo received at least one dose of aprocitentan 25 mg during part 3.) | 0 | 0 | 0 | 0 | 310 | 303
Completed | 0 | 0 | 0 | 0 | 288 | 289
Not Completed | 0 | 0 | 0 | 0 | 19 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 8 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons | 0 | 0 | 0 | 0 | 9 | 6
Not completed — Re-randomized in part 3, however no drug dispensed | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aprocitentan 12.5 mg in Part 1 (Double-blind): Participants randomized to aprocitentan 12.5 mg, orally, once daily in the morning for 4 weeks.
- Aprocitentan 25 mg in Part 1 (Double-blind): Participants randomized to aprocitentan 25 mg, orally, once daily in the morning for 4 weeks.
- Placebo in Part 1 (Double-blind): Participants randomized to placebo (matching aprocitentan), orally, once daily in the morning for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind) | Total
Number analyzed (Participants) | 243 | 243 | 244 | 730
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.3) | 61.7 (10.4) | 62.2 (11.2) | 61.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 99 | 296
  Male | 144 | 145 | 145 | 434
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 22 | 23 | 73
  Not Hispanic or Latino | 213 | 219 | 218 | 650
  Unknown or Not Reported | 2 | 2 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 14 | 13 | 38
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 28 | 28 | 26 | 82
  White | 203 | 200 | 202 | 605
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 8 | 7 | 23
  Belgium | 1 | 3 | 4 | 8
  Canada | 8 | 7 | 6 | 21
  China | 6 | 11 | 10 | 27
  Czechia | 10 | 3 | 15 | 28
  Finland | 9 | 5 | 2 | 16
  France | 0 | 4 | 3 | 7
  Germany | 3 | 6 | 9 | 18
  Greece | 5 | 1 | 2 | 8
  Hungary | 1 | 4 | 1 | 6
  Israel | 5 | 2 | 3 | 10
  Italy | 3 | 2 | 0 | 5
  Lithuania | 2 | 4 | 4 | 10
  Netherlands | 2 | 3 | 3 | 8
  Poland | 15 | 16 | 20 | 51
  Russia | 61 | 56 | 49 | 166
  Spain | 4 | 8 | 6 | 18
  Ukraine | 30 | 26 | 30 | 86
  United Kingdom | 2 | 0 | 1 | 3
  United States | 68 | 74 | 69 | 211
Body Mass Index at Screening Visit [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (6.2) | 34.3 (6.8) | 33.3 (5.6) | 33.7 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 of Double-blind Treatment in Mean Trough Sitting Systolic Blood Pressure (SiSBP) Measured by Automated Office Blood Pressure Measurement
Description: Changes from baseline to Week 4 in mean trough SiSBP were analyzed using a mixed model. Participants had their blood pressure (BP) measured at the study site using the automated oscillometric sphygmomanometer (Microlife WatchBP® Office) which was provided to each site. BP was to be measured at trough (before taking the study treatment and SBAT). The BP assessment, participant preparation (e.g., arm selection, arm position, cuff size) was standardized and followed the American Heart Association guidelines / Canadian Education Program on Hypertension. The participant was resting undisturbed, alone (unattended) in a quiet place for 5 minutes at each visit. BP was measured at each visit with the same device, which recorded five sitting blood pressure readings (one per minute, the first value was excluded from the average). A negative change indicates a decrease in SiSBP from baseline.
Time Frame: Pre-dose Day 1 (Part 1 double-blind randomized baseline) up to Week 4 (End of double-blind randomized part 1)
Population: The Full Analysis Set (FAS) includes all participants who were randomized and had a baseline sitting systolic blood pressure, measured by automated office blood pressure measurement. Baseline was defined as the last measurement before randomization.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: mmHg
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind)
Number analyzed (Participants) | 243 | 243 | 244
mmHg | -15.26 [-17.36 to -13.17] | -15.20 [-17.27 to -13.13] | -11.47 [-13.57 to -9.38]
Statistical Analysis 1: Comparison: Aprocitentan 12.5 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); Test type: Superiority; p = 0.0042, Mixed Models Analysis — Mixed effects model for Repeated Measures: Change from baseline in SiSBP = baseline SiSBP + treatment + visit + treatment x visit + baseline x visit; LS Mean difference to placebo = -3.79, 97.5% CI 2-sided [-6.76 to -0.82]
Statistical Analysis 2: Comparison: Aprocitentan 25 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); Test type: Superiority; p = 0.0046, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean difference to placebo = -3.73, 97.5% CI 2-sided [-6.67 to -0.78]

2. Secondary Outcome: Change From Double-blind Withdrawal Baseline (Week 36) to Week 40 in Mean Trough Sitting Systolic Blood Pressure (SiSBP) Measured by Unattended Automated Office Blood Pressure Measurement
Description: Changes from double-blind withdrawal baseline (Week 36) to Week 40 in mean trough SiSBP were analyzed using a mixed model. Participants had their blood pressure (BP) measured at the study site using the automated oscillometric sphygmomanometer (Microlife WatchBP® Office) which was provided to each site. BP was to be measured at trough (before taking the study treatment and SBAT). The BP assessment, participant preparation (e.g., arm selection, arm position, cuff size) was standardized and followed the American Heart Association guidelines / Canadian Education Program on Hypertension. The participant was resting undisturbed, alone (unattended) in a quiet place for 5 minutes at each visit. BP was measured at each visit with the same device, which recorded five sitting blood pressure readings (one per minute, the first value was excluded from the average). A negative change indicates a decrease in SiSBP from baseline.
Time Frame: Pre-dose Week 36 (Part 3 double-blind-withdrawal baseline) up to Week 40
Population: The modified FAS (mFAS) includes all participants from the FAS who were re-randomized in the double-blind-withdrawal part (DB-WD) of the study and who have a DB-WD baseline sitting systolic blood pressure, measured by automatic office blood pressure measurement device at trough. Baseline was defined as the last measurement before re-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal): After 32-weeks in the single-blind, single-arm part, participants were re-randomized to aprocitentan 25 mg, orally, once daily in the morning for 12 weeks.
- Placebo in Part 3 (Double-blind Withdrawal): After 32-weeks in the single-blind, single-arm part, participants were re-randomized to placebo (matching aprocitentan), orally, once daily in the morning for 12 weeks.
Arm/Group | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Number analyzed (Participants) | 307 | 307
mmHg | -1.47 [-2.97 to 0.04] | 4.36 [2.87 to 5.85]
Statistical Analysis 1: Comparison: Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) vs Placebo in Part 3 (Double-blind Withdrawal); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Mixed effects model for Repeated Measures: Change from DB-WD baseline in SiSBP = DB-WD baseline SiSBP + stratum (randomized treatment in DB part) + treatment + visit + treatment x visit + DB-WD baseline x visit; LS mean difference to placebo. = -5.82, 95% CI 2-sided [-7.94 to -3.71]

3. Secondary Outcome: Change From Baseline to Week 4 of Double-blind Treatment in Mean Trough Sitting Diastolic Blood Pressure (SiDBP) Measured by Unattended Automated Office Blood Pressure Measurement
Description: Changes from baseline to Week 4 in mean trough SiDBP were analyzed using a mixed model. Participants had their blood pressure (BP) measured at the study site using the automated oscillometric sphygmomanometer (Microlife WatchBP® Office) which was provided to each site. BP was to be measured at trough (before taking the study treatment and SBAT). The BP assessment, participant preparation (e.g., arm selection, arm position, cuff size) was standardized and followed the American Heart Association guidelines / Canadian Education Program on Hypertension. BP was measured at each visit with the same device, which recorded five sitting blood pressure readings (one per minute, the first value was excluded from the average). The participant was resting undisturbed, alone (unattended) in a quiet place for 5 minutes at each visit. A negative change indicates a decrease in SiDBP from baseline.
Time Frame: Pre-dose Day 1 (Part 1 double-blind randomized baseline) up to Week 4 (End of double-blind randomized part 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind)
Number analyzed (Participants) | 243 | 243 | 244
mmHg | -10.43 [-11.58 to -9.27] | -10.95 [-12.09 to -9.82] | -6.48 [-7.63 to -5.33]
Statistical Analysis 1: Comparison: Aprocitentan 12.5 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); Test type: Other; p < 0.0001, Mixed Models Analysis — Mixed effects model for Repeated Measures: Change from baseline in SiDBP = baseline SiDBP + treatment + visit + treatment x visit + baseline x visit; LS Mean difference to placebo = -3.94, 95% CI 2-sided [-5.57 to -2.31]
Statistical Analysis 2: Comparison: Aprocitentan 25 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; LS Mean difference to placebo = -4.47, 95% CI 2-sided [-6.09 to -2.85]

4. Secondary Outcome: Changes From Baseline to Week 4 of Double-blind Treatment in 24-hour Mean Systolic (SBP) and Diastolic Blood Pressure (DBP) Measured by Ambulatory Blood Pressure Monitoring
Description: ABPM devices were provided to each site by the central blood pressure laboratory. On the first day after all visit assessments were performed, the ABPM device (Mobil-O-Graph NG) was fitted to the participant. The following day (i.e., second day), the participant came back to site to have the ABPM device removed. ABPM data collected over the 24-hours was electronically transferred to the central BP laboratory. Systolic blood pressure and diastolic blood pressure were measured at predetermined times every 20 minutes from 06:00 to 21:59, and every 30 minutes from 22:00 to 05:59. For each participant and at each visit (baseline and Week 4) the 24-hour mean SBP (or DBP) was calculated from the area under the SBP (or DBP) time curve and divided by the time span. A negative change indicates a decrease in 24-hour mean systolic / diastolic blood pressure from baseline.
Time Frame: Pre-dose Day 1 (Part 1 double-blind randomized baseline) and Week 4 (End of double-blind randomized part 1)
Population: The ambulatory blood pressure monitoring full analysis set (aFAS) includes all participants from the FAS who have a baseline 24-hour mean systolic and diastolic blood pressure measured by ambulatory blood pressure monitoring with a total duration of at least 21 hours and at least 70% valid readings.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind)
Number analyzed (Participants) | 206 | 207 | 220
mmHg
  24-hour mean systolic blood pressure | -6.73 [-8.20 to -5.26] | -8.44 [-9.88 to -7.00] | -2.55 [-4.00 to -1.10]
  24-hour mean diastolic blood pressure | -6.25 [-7.20 to -5.29] | -7.74 [-8.67 to -6.80] | -1.92 [-2.87 to -0.98]
Statistical Analysis 1: Comparison: Aprocitentan 12.5 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); 24-hour mean systolic (SBP); Test type: Other; p < 0.0001, ANCOVA; LS Mean difference to placebo = -4.18, 95% CI 2-sided [-6.25 to -2.12]
Statistical Analysis 2: Comparison: Aprocitentan 25 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); 24-hour mean systolic (SBP); Test type: Other; p < 0.0001, ANCOVA; LS Mean difference to placebo = -5.90, 95% CI 2-sided [-7.94 to -3.85]
Statistical Analysis 3: Comparison: Aprocitentan 12.5 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); 24-hour mean diastolic (DBP); Test type: Other; p < 0.0001, ANCOVA; LS Mean difference to placebo = -4.32, 95% CI 2-sided [-5.66 to -2.98]
Statistical Analysis 4: Comparison: Aprocitentan 25 mg in Part 1 (Double-blind) vs Placebo in Part 1 (Double-blind); 24-hour mean diastolic (DBP); Test type: Other; p < 0.0001, ANCOVA; LS Mean = -5.81, 95% CI 2-sided [-7.14 to -4.49]

5. Secondary Outcome: Change From Double-blind Withdrawal Baseline (Week 36) to Week 40 of Double-blind-withdrawal (DB-WD) Treatment in Trough Sitting Diastolic Blood Pressure (SiDBP) Measured by Unattended Automated Office Blood Pressure
Description: Changes from double-blind withdrawal (Week 36) to Week 40 in mean trough SiDBP were analyzed using a mixed model. Participants had their blood pressure (BP) measured at the study site using the automated oscillometric sphygmomanometer (Microlife WatchBP® Office) which was provided to each site. BP was to be measured at trough (before taking the study treatment and SBAT). The BP assessment, participant preparation (e.g., arm selection, arm position, cuff size) was standardized and followed the American Heart Association guidelines / Canadian Education Program on Hypertension. The participant was resting undisturbed, alone (unattended) in a quiet place for 5 minutes at each visit. BP was measured at each visit with the same device, which recorded five sitting blood pressure readings (one per minute, the first value was excluded from the average). A negative change indicates a decrease in SiDBP from baseline.
Time Frame: Pre-dose Week 36 (Part 3 double-blind-withdrawal baseline) up to Week 40
Population: The modified FAS (mFAS) includes all participants in the FAS who were re-randomized in the double-blind-withdraw part of the study and who had a week 36 sitting systolic blood pressure, measured by automated office blood pressure measurement. Baseline was defined as the last measurement before re-randomization into part 3 of the double-blind withdrawal part of the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Number analyzed (Participants) | 307 | 307
mmHg | -0.52 [-1.54 to 0.50] | 4.67 [3.66 to 5.68]
Statistical Analysis 1: Comparison: Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) vs Placebo in Part 3 (Double-blind Withdrawal); Test type: Other; p < 0.0001, Mixed Models Analysis — Mixed effects model for Repeated Measures: Change from DB-WD baseline in SiDBP = Double-blind withdrawal baseline SiDBP + stratum (randomized treatment in DB part) + treatment + visit + treatment x visit + Double-blind withdrawal baseline x visit; LS Mean difference to placebo = -5.19, 95% CI 2-sided [-6.62 to -3.76]

6. Secondary Outcome: Changes From Double-blind Withdrawal Baseline (Week 36) to Week 40 of Double-blind-withdrawal (DB-WD) Treatment in 24-hour Mean Systolic (SBP) and Diastolic Blood Pressure (DBP) Measured by Ambulatory Blood Pressure Monitoring
Description: ABPM devices were provided to each site by the central blood pressure laboratory. On the first day after all visit assessments were performed, the ABPM device (Mobil-O-Graph NG) was fitted to the participant. The following day (i.e., second day), the participant came back to site to have the ABPM device removed. ABPM data collected over the 24-hours was electronically transferred to the central BP laboratory. Systolic blood pressure and diastolic blood pressure were measured at predetermined times every 20 minutes from 06:00 to 21:59, and every 30 minutes from 22:00 to 05:59. For each participant and at each visit (the double-blind withdrawal baseline [Week 36] and the week 40) the 24-hour mean SBP (or DBP) was calculated from the area under the SBP (or DBP) time curve. A negative change indicates a decrease in 24-hour mean systolic / diastolic blood pressure from baseline.
Time Frame: From Week 36 (Part 3 double-blind-withdrawal baseline) and Week 40
Population: The modified ambulatory blood pressure monitoring full analysis set (maFAS) includes all participants from the modified Full Analysis Set (mFAS) who had a double-blind withdrawal (DB-WD) baseline 24-hour mean systolic and diastolic blood pressure, measured by ambulatory blood Pressure monitoring (ABPM) with a total duration of at least 21 hours and at least 70% valid readings.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
Number analyzed (Participants) | 237 | 241
mmHg
  24-hour mean systolic blood pressure | -0.07 [-1.46 to 1.32] | 6.46 [5.06 to 7.85]
  24-hour mean diastolic blood pressure | -0.47 [-1.34 to 0.40] | 6.28 [5.40 to 7.15]
Statistical Analysis 1: Comparison: Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) vs Placebo in Part 3 (Double-blind Withdrawal); 24-hour mean systolic (SBP); Test type: Other; p < 0.0001, ANCOVA; LS Mean difference to placebo = -6.53, 95% CI 2-sided [-8.50 to -4.56]
Statistical Analysis 2: Comparison: Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) vs Placebo in Part 3 (Double-blind Withdrawal); 24-hour mean diastolic (DBP); Test type: Other; p < 0.0001, ANCOVA; LSM Mean difference to placebo = -6.75, 95% CI 2-sided [-7.98 to -5.52]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment-emergent, if the onset date is between the first intake of treatment up to 30 days after the stop of study treatment. Study treatment was for up to 48 weeks. In Part 1 double-blind (DB) treatment was for 4 weeks. Part 2 single-blind (SB) study treatment was for 32 weeks. In Part 3 double-blind withdrawal (DB-WD) study treatment was for 12 weeks.
Description: Only participants entering the randomized treatment period were considered enrolled for the study and are included in AE analysis. The Run-in period was designed to exclude potential placebo responders and is not part of statistical analysis of this study.
Groups:
- Aprocitentan 12.5 mg in Part 1 (Double-blind): Participants received aprocitentan 12.5 mg, orally, once daily in the morning for 4 weeks.
- Aprocitentan 25 mg in Part 1 (Double-blind): Participants received aprocitentan 25 mg, orally, once daily in the morning for 4 weeks.
- Placebo in Part 1 (Double-blind): Participants received placebo, orally, once daily in the morning for 4 weeks.
- Aprocitentan 25 mg in Part 2 (Single-blind): All participants received aprocitentan 25 mg, orally, once daily in the morning for 32 weeks.
- Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal): After 32-weeks in the single-blind, single-arm part, participants received aprocitentan 25 mg, orally, once daily in the morning for 12 weeks.
- Placebo in Part 3 (Double-blind Withdrawal): After 32-weeks in the single-blind, single-arm part, participants received placebo (matching aprocitentan), orally, once daily in the morning for 12 weeks.
Arm/Group | Aprocitentan 12.5 mg in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 1 (Double-blind) | Placebo in Part 1 (Double-blind) | Aprocitentan 25 mg in Part 2 (Single-blind) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) | Placebo in Part 3 (Double-blind Withdrawal)
All-Cause Mortality (participants affected / at risk) | 1/243 | 0/245 | 0/242 | 9/704 | 1/310 | 0/303
Serious Adverse Events (participants affected / at risk) | 8/243 | 8/245 | 3/242 | 82/704 | 18/310 | 9/303
Other Adverse Events (participants affected / at risk) | 16/243 | 34/245 | 5/242 | 95/704 | 6/310 | 4/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprocitentan 12.5 mg in Part 1 (Double-blind) (N=243) | Aprocitentan 25 mg in Part 1 (Double-blind) (N=245) | Placebo in Part 1 (Double-blind) (N=242) | Aprocitentan 25 mg in Part 2 (Single-blind) (N=704) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) (N=310) | Placebo in Part 3 (Double-blind Withdrawal) (N=303)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 14 (14) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprocitentan 12.5 mg in Part 1 (Double-blind) (N=243) | Aprocitentan 25 mg in Part 1 (Double-blind) (N=245) | Placebo in Part 1 (Double-blind) (N=242) | Aprocitentan 25 mg in Part 2 (Single-blind) (N=704) | Aprocitentan 25 mg in Part 3 (Double-blind Withdrawal) (N=310) | Placebo in Part 3 (Double-blind Withdrawal) (N=303)
Oedema peripheral (General disorders) | 16 (16) | 34 (34) | 5 (5) | 95 (102) | 6 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (3):
  • Study Protocol: Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03541174/Prot_000.pdf
  • Study Protocol: Protocol Addendum Covid-19 (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT03541174/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03541174/SAP_002.pdf